CLINICAL TRIAL: NCT04563689
Title: Efecto de un Enjuague Bucal Con Clorhexidina al 0.12% y Cloruro de Cetil Piridinio al 0.05% en la Carga Viral en Saliva en Pacientes COVID-19 + Hospitalizados o Que Esten Recibiendo Cuidado médico en Casa en Cali - 2020.
Brief Title: Pilot Study to Evaluate Effect of CHX0.12/CPC 0.05 of SARS-CoV-2 Viral Load in COVID-19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dentaid SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: COVID-POC1
Record Dates: First submitted 2020-09-22; First posted 2020-09-24 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- actve (Experimental): oral rinse
  Interventions: Other: CHX0.12+CPC0.05 oral rinse (PerioAidActive Control)
- placebo (Placebo Comparator): distilled water,
  Interventions: Other: placebo rinse

INTERVENTIONS:
Other: CHX0.12+CPC0.05 oral rinse (PerioAidActive Control) — rinse 15 ml during 1 min during 5 days, twice daily
  Arms: actve
Other: placebo rinse — destilled water rinse 15 ml during 1 min during 5 days, twice daily
  Arms: placebo

SUMMARY:
Randomized, double-blind, placebo-controlled pilot study to evalaute viral load in saliva of COVID19+ patients using quantitative PCR, before and after use of active or placebo rinses

ELIGIBILITY:
Inclusion Criteria:

1. Be positive for SARS-CoCV-2 real-time PCR test
2. SARS-CoV-2 patients positive, with home and/or hospitalized care.
3. Have a medical condition that allows them to perform a mouthwash for 1 minute.

Exclusion Criteria:

1. Pregnant.
2. People with impaired lung function who do not allow them to rinse.
3. Patients with antiviral treatment for Covid-19.
4. Patients with diseases that affect saliva, Sjogren's syndrome, and Systemic Lupus Erythematosus.
5. Any cause of immunosuppression (primary or secondary), including HIV.
6. Chronic kidney disease 3b or older, Coronary heart disease, Uncontrolled diabetes (Hb1Ac >7), Uncontrolled high blood pressure, Uncontrolled thyroid disease, history of cancer less than 1 year

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2020-10-22 (Actual); Study Completion 2020-10-23 (Actual)

PRIMARY OUTCOMES:
exploratory change in viral load | baseline (pre-rinse) and 15 min, 1 hour, 2 hours and 5 days after initial oral rinse
  change versus baseline in viral load of SARS-CoV-2 in spontaneous saliva measured by quantitative PCR

SECONDARY OUTCOMES:
number of patients who have decrease in viral load of SARS-CoV-2 in spontaneous saliva measured by quantitative PCR | 15 min, 1 hour, 2 hours and 5 days after initial oral rinse
  number of patients who have decrease in viral load of SARS-CoV-2 in spontaneous saliva measured by quantitative PCR
number of patients with adverse events during 5 days study duration | through study completion in day 5
  description of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Leon, PhD, Study Director — Dentaid SL
Locations (1):
- Escuela odontologia. Facultad de Salud Hospital del Valle, Cali, Colombia